CLINICAL TRIAL: NCT07022262
Title: 3D-BONE: Virtual Exercise Training and Its Impact on Cortical and Trabecular Bone Compartments in Adult Survivors of Childhood Cancer: a Peripheral Quantitative Computed Tomography (pQCT) Study
Brief Title: Virtual Exercise Training and Its Impact on Bone Compartments in Adult Survivors of Childhood Cancer
Acronym: 3D-BONE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Loyola University (Other); University of Thessaly (Other); Hospital Materno-Infantil Torrecárdenas de Almería (Unknown); Hospital Universitario Reina Sofia de Cordoba (Other Government); University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Esther Ubago Guisado, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Universidad de Granada; PID2023-150311OB-I00 (Other Grant/Funding Number: Ministerio de Ciencia, Innovación y Universidades)
Record Dates: First submitted 2025-05-26; First posted 2025-06-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cancer Survivors
Keywords: cancer survivors; childhood cancer; exercise; bone health; physical fitness; sarcopenia; physiological frailty; mental health; health-related quality of life; pQCT
MeSH Terms: conditions — Neoplasms; Motor Activity; Sarcopenia; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 6-months of live and online progressive resistance training plus impact loading + dietary counselling on calcium and vitamin D.
  Interventions: Behavioral: Progressive resistance training plus impact loading
- Control group (No Intervention): Dietary counselling on calcium and vitamin D.

INTERVENTIONS:
Behavioral: Progressive resistance training plus impact loading — The structure of the exercise sessions will be: 1) warm up; 2) progressive resistance training plus impact loading; 3) cool down. Briefly, the warm-ups will be based on RAMP methodology (i.e., raise, activate, mobilise and potentiate) in order to maximize middle-term performance of the main exercises. Exercises focused on the brace, squat, lunge or jump patterns will be included in the first part of the session. The main part of the session will consist of 9 sets of 10-12 jumps, 9 sets of 10-12 repetitions of lower body resistance exercise and 3 sets of 10-12 repetitions of upper resistance exercise. Each set will be performed with approximately 15-30 seconds of rest for jumps and 2-3 minutes of rest for resistance exercises. Finally, participants will perform a cool down including guided static stretching and relaxing exercises.
  Arms: Intervention group

SUMMARY:
Childhood cancer is a rare disease but a significant cause of death in children and adolescents. The incidence of childhood cancer is 1case per 300 cases of adult cancer, but surviving to it has important sequels. Endocrine dysfunction represents one of the most common issues in paediatric cancer survivors and impairs bone mineral density later in life. Some forms of exercise have been recommended to preserve bone health in healthy adults; however, its effect has not been properly studied yet in adult survivors of paediatric cancer using cutting-edge technologies, such as peripheral quantitative computed tomography (pQCT). As general aim, the 3D-BONE study will assess for the first time the effect of a live and online exercise programme on bone parameters and bone metabolism in adult survivors of paediatric cancer. This multicenter randomized controlled trial will be performed in three Andalusian provinces (Granada, Cordoba and Almeria). A minimum of 116 adult survivors of paediatric cancer aged 18 to 55 years will be recruited following the inclusion and exclusion criteria. They will be randomized (based on sex and age) into an INTERVENTION (n=58) or CONTROL group (n=58). The intervention group will receive a 6-month live and online exercise program based on progressive resistance and impact loading training that will be delivered by qualified professionals using a telehealth mobile app (3D-BONE app). Moreover, behaviour change techniques will be implemented in order to increase motivation and adherence to the program. This group will also receive diet counselling on calcium and vitamin so the difference between the groups is the exercise programme. Participants will be assessed before and after the intervention at the facilities of the Sport and Health University Research Institute (iMUDS) of the University of Granada. An in-depth analysis of bone parameters will be carried out using cutting-edge technologies, such as the pQCT (to analyse cortical and trabecular bone in 3 dimensions), dual-energy X-ray absorptiometry (DXA), hip and lumbar spine geometry outcomes. Moreover, a complete blood count will be obtained and markers of bone metabolism will be measured (B-CTX, PINP), including novel markers such as sclerostin and irisin which have recently been linked to human bone. Data will also be collected in anthropometry and body composition to obtain cardiovascular risk factors, sarcopenia and physiologic frailty risk factors, mental health, health-related quality of life and objective measures of physical activity and fitness. This will ensure obtaining novel, precise and strong data in this population.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of pediatric cancer and history of receiving treatment (radiation therapy and/or chemotherapy).
* 18-55 years of age at recruitment

Exclusion Criteria:

* Participation in another research study simultaneously.
* Not currently receiving cancer treatment.
* Previous diagnosed anorexia/bulimia, known pregnancy, known alcohol or drug abuse.
* Requiring chronic oral glucocorticoid therapy.
* Having an injury that may affect daily life activities and can be aggravated by exercise.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Cortical and Trabecular Volumetric Bone Mineral Density (pQCT) | Baseline and 6 months
  Cortical and trabecular BMD will be measured at tibia and radius using pQCT (mg/cm³).
Change in Cortical Bone Thickness (pQCT) | Baseline and 6 months
  Cortical bone thickness at tibia and radius (mm) will be derived from pQCT images.
Change in Periosteal and Endocortical Circumference (pQCT) | Baseline and 6 months
  Periosteal and endocortical circumference at tibia and radius will be measured via pQCT (mm)
Change in Cross-Sectional Moment of Inertia-CSMI (pQCT) | Baseline and 6 months
  CSMI at tibia and radius will be calculated to assess structural bone strength (mm⁴).
Change in Muscle Area (pQCT) | Baseline and 6 months
  Muscle area at tibia and radius will be obtained from pQCT images (cm²)
Change in Bone Mineral Content (DXA) | Baseline and 6 months
  BMC will be assessed using DXA at whole-body and regional sites (g)
Change in Areal Bone Mineral Density (DXA) | Baseline and 6 months
  Areal BMD will be measured with DXA at whole-body and regional sites (g/cm²)
Change in Cross-Sectional Area (DXA-HSA) | Baseline and 6 months
  Derived from hip structural analysis (mm²).
Change in Section Modulus (DXA-HSA) | Baseline and 6 months
  Indicates bone strength; calculated from HSA (mm³).
Change in Cross-Sectional Moment of Inertia (DXA-HSA) | Baseline and 6 months
  Assesses resistance to bending forces (mm⁴).
Change in Trabecular Bone Score (TBS) | Baseline and 6 months
  Lumbar spine texture will be assessed using TBS (TBS index).
Change in Serum Lipid Profile | Baseline and 6 months
  Cholesterol, triglycerides, HDL, LDL levels (mg/dL).
Change in Total bilirubin | Baseline and 6 months
  mg/dL
Change in Calcium | Baseline and 6 months
  mg/dL
Change in Creatinine | Baseline and 6 months
  mg/dL
Change in Phosphorus | Baseline and 6 months
  mg/dL
Change in Glucose | Baseline and 6 months
  mg/dL
Change in Magnesium | Baseline and 6 months
  mg/dL
Change in Uric acid | Baseline and 6 months
  mg/dL
Change in ALT/GPT | Baseline and 6 months
  U/L
Change in Na/K/Cl | Baseline and 6 months
  mEq/L
Change in Albumin | Baseline and 6 months
  g/dL
Change in Total protein | Baseline and 6 months
  g/dL
Change in Serum 25(OH) Vitamin D | Baseline and 6 months
  ng/mL
Change in Alkaline phosphatase | Baseline and 6 months
  U/L
Change in Bone specific alkaline phosphatase | Baseline and 6 months
  ng/mL
Change in Glycosylated hemoglobin | Baseline and 6 months
  mmol/mol
Change in Parathyrin | Baseline and 6 months
  pg/mL
Change in Thyrotropin | Baseline and 6 months
  µUI/mL
Change in Gamma-glutamyl transferase | Baseline and 6 months
  U/L
Change in β-CTX (Serum) | Baseline and 6 months
  Marker of bone resorption (ng/mL)
Change in PINP (Serum) | Baseline and 6 months
  Marker of bone formation (ng/mL)
Change in Irisin (Serum) | Baseline and 6 months
  ng/mL
Change in Sclerostin (Serum) | Baseline and 6 months
  ng/mL

SECONDARY OUTCOMES:
Change in Body Mass | Baseline and 6 months
  Measured with electronic scale (kg).
Change in Height | Baseline and 6 months
  Measured with stadiometer (cm).
Change in Body Mass Index (BMI) | Baseline and 6 months
  Calculated as kg/m².
Change in Blood Pressure | Baseline and 6 months
  Systolic and diastolic pressure measured in mmHg.
Change in body circumferences | Baseline and 6 months
  Waist, hip and neck circumferences measured in cm.
Change in Lean Soft Tissue Mass (DXA) | Baseline and 6 months
  Assessed at whole-body using DXA (g).
Change in Fat Mass (DXA) | Baseline and 6 months
  Assessed at whole-body using DXA (kg).
Change in Body Fat Percentage (DXA) | Baseline and 6 months
  Assessed at whole-body using DXA (%).
Change in 6-Minute Walk Test | Baseline and 6 months
  Distance walked in 6 minutes (meters).
Change in Squat Jump Test | Baseline and 6 months
  Height achieved in the test (cm).
Change in Handgrip Strength Test | Baseline and 6 months
  Maximal grip force (kg).
Change in Standing Long Jump Test | Baseline and 6 months
  Distance achieved in the test (cm).
Change in 5 Times Sit-to-Stand Test | Baseline and 6 months
  Time to complete 5 repetitions (seconds)
Change in 4-m Gait Speed Test | Baseline and 6 months
  Time to walk 4 meters (seconds)
Change in Self-Reported Fitness (IFIS) | Baseline and 6 months
  Perceived fitness using IFIS questionnaire.
Change in Sarcopenia Classification (EWGSOP2) | Baseline and 6 months
  Sarcopenia will be classified as no, probable, or confirmed based on grip strength, sit-to-stand time, and appendicular lean mass by DXA. Categorical (no/probable/confirmed).
Change in Frailty Status | Baseline and 6 months
  Frailty will be assessed using five criteria: low muscle mass, fatigue, low physical activity, slowness, and weakness. Categorical (frail/non-frail).
Change in Physical Activity and Sedentarism (Accelerometer) | Baseline and 6 months
  Measured over 7 consecutive days using ActiGraph (counts per minute).
Change in Self-Reported Physical Activity (IPAQ) | Baseline and 6 months
  Activity levels using the IPAQ (MET-min/week)
Change in Bone-Specific Physical Activity (BPAQ) | Baseline and 6 months
  Scored from the BPAQ questionnaire (BPAQ score)
Change in Calcium Intake | Baseline and 6 months
  Estimated using validated short calcium questionnaire (mg/day).
Change in Vitamin D Intake | Baseline and 6 months
  Estimated from dietary questionnaire (IU/day).
Change in Mediterranean Diet Adherence | Baseline and 6 months
  Calculated from validated adherence questionnaire (Score 0-14)
Change in Quality of Life | Baseline and 6 months
  HRQoL from the SF-36 questionnaire (0-100 scale).
Change in Anxiety and Depression (HADS) | Baseline and 6 months
  Anxiety and depression score from HADS (Score 0-21)
Change in Self-Esteem (Rosenberg Scale) | Baseline and 6 months
  Assessed using Rosenberg Self-Esteem Scale (Score 0-30)
Change in Perceived Stress (PSS) | Baseline and 6 months
  Assessed via Perceived Stress Scale (Score 0-40).

OTHER OUTCOMES:
Change in objective strength | Baseline and 6 months
  Objective strength will be measured with a functional electromechanical dynamometer-DynaSystem (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Health University Research Institute (iMUDS), Technological Health Park, University of Granada, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data files including IPD and corresponding data dictionaries will be shared under restricted access and upon reasonable request (E Ubago-Guisado or L Gracia-Marco) due to privacy issue and GDPR regulations. In principle, all collected IPD will be available for sharing under the "as open as possible, as closed as necessary" principle. The shared data files will be pseudonymized, only include participants who provided informed consent for sharing, and sharing is only possible when the data is used for research purposes. This is stated at the informed consent files that the participants signed when they agree to participate.